CLINICAL TRIAL: NCT02936362
Title: Testing the Effect of Whole-wheat Sourdough Bread Compared to White Bread on Healthy Individuals: Randomized Trial
Brief Title: Testing the Effect of Whole-wheat Sourdough Bread Compared to White Bread on Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-12-ZH-658A
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Dietary Modification; Bread; Gastrointestinal Microbiome; Hematologic Tests; Body Weight Changes
Keywords: Bread; Microbiome; Blood tests; Sourdough bread; Dietary intervention
MeSH Terms: conditions — Body Weight Changes

ARMS (2):
- Sourdough bread, white bread (Other): Consumption of sourdough bread for one week, 2 week washout, consumption of white bread for one week
  Interventions: Other: Consumption of sourdough bread; Other: Consumption of white bread
- White bread, sourdough bread (Other): Consumption of white bread for one week, 2 week washout, consumption of sourdough bread for one week
  Interventions: Other: Consumption of sourdough bread; Other: Consumption of white bread

INTERVENTIONS:
Other: Consumption of sourdough bread — Participants will be given sourdough bread to consume instead of other wheat products. 145g will be consumed every morning in addition to ad libitum consumption throughout the day (matched between first and second intervention periods)
Other: Consumption of white bread — Participants will be given white bread to consume instead of other wheat products. 110g will be consumed every morning in addition to ad libitum consumption throughout the day (matched between first and second intervention periods)

SUMMARY:
Bread is the most common grain product in the world, with consumption surpassing 3 billion individuals per year. Sourdough whole-grain bread is considered a healthy alternative to white, refined-wheat bread.

This cross-over study will test the effect of consumption of sourdough bread compared to white bread following a short dietary intervention period (one week) on multiple clinical parameters and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide and signed informed consent form
* Over 18 years
* Not in active military service
* Ability to technically operate a glucometer

Exclusion Criteria:

* Prediagnosed type I / type II diabetes mellitus
* Pregnancy
* Usage of antibiotics within three months prior to participation
* Chronically active inflammatory or neoplastic disease in the three years prior to enrollment
* Skin disease, including contact dermatitis, precluding proper attachment of the continuous glucose monitor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes to glycemic control | One week
  Measured as response to an Oral Glucose Tolerance Test (OGTT; mg/dl*h).
Changes to glycemic control | One week
  Measured as blood glucose levels at wake-up (mg/dl).

SECONDARY OUTCOMES:
Changes to total cholesterol levels (mg/dl) | One week
  Measured by a blood test.
Changes to HDL cholesterol levels (mg/dl) | One week
  Measured by a blood test.
Changes to LDL cholesterol levels (mg/dl) | One week
  Measured by a blood test.
Changes to triglycerides levels (mg/dl) | One week
  Measured by a blood test.
Changes to C-Reactive Protein (CRP) levels (mg/l) | One week
  Measured by a blood test.
Changes to weight (Kg.) | One week
Changes to Basal Metabolic Rate (BMR; J) | One week
Changes to blood pressure (mmHg) | One week
Changes to Alanine Transaminase (ALT) levels (IU/l) | One week
  Measured by a blood test.
Changes to Aspartate Transaminase (AST) levels (IU/I) | One week
  Measured by a blood test.
Changes to Gamma-Glutamyl Transpeptidase (GGT) levels (IU/l) | One week
  Measured by a blood test.
Changes to Creatinine levels (mg/dl) | One week
  Measured by a blood test.
Changes to Magnesium levels (mg/dl) | One week
  Measured by a blood test.
Changes to Calcium levels (mg/dl) | One week
  Measured by a blood test.
Changes to Iron levels (mg/dl) | One week
  Measured by a blood test.
Changes to Urea levels (mg/dl) | One week
  Measured by a blood test.
Changes to Lactate Dehydrogenase (LDH) levels | One week
  Measured by a blood test (IU/l)
Changes to Thyroid Stimulating Hormone (TSH) | One week D
  Measured by a blood test (mIU/ml)

OTHER OUTCOMES:
Changes to gut microbiome composition and function | One week
  Measured by metagenomic sequencing

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Weizmann Institute of Science, Rehovot
  - Department of Gastroentherology, Tel Aviv